CLINICAL TRIAL: NCT00319813
Title: General Practice Quality Assurance Project. COPD Diagnosis and Treatment
Brief Title: General Practice Quality Assurance Project. Chronic Obstructive Pulmonary Disease (COPD) Diagnosis and Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.376; NCT00479869 (obsolete NCT alias)
Record Dates: First submitted 2006-04-20; First posted 2006-04-27 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education

SUMMARY:
A Cross sectional observational Quality Assurance Project in General Practice to COPD Diagnosis and Treatment

ELIGIBILITY:
Inclusion Criteria:

* COPD patients over 35 years of age
* More than two annual renewals with the following group of inhalation preparations: Anticholinergic, beta-2 antagonists, steroids or a combination of these

Exclusion Criteria:

* Asthma

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 2006-04-19 (Actual); Primary Completion 2007-09-05 (Actual); Study Completion 2007-09-05 (Actual)

PRIMARY OUTCOMES:
To optimise the diagnosis and treatment of COPD via a quality assurance project | Up to 1.2 years
Increase the knowledge and use of diagnostic tools and treatment amongst PCPs | Up to 1.2 years
To focus on implementation of national guidelines for diagnosis and treatment of COPD | Up to 1.2 years

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Denmark A/S